CLINICAL TRIAL: NCT01645345
Title: RF Pixel With Micro-Plasma Technology: Fractional Ablative Radiofrequency for the Treatment of Acne Scars and RF Pixel With Micro-Plasma Technology: Fractional Ablative Radiofrequency for the Treatment of Acne Scars and
Brief Title: Fractional Ablative Radiofrequency for the Treatment of Acne Scars and Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alma Lasers Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 022012
Record Dates: First submitted 2012-07-13; First posted 2012-07-20 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2012-07

CONDITIONS: Wrinkles; Acne Scars
Keywords: wrinkles; acne scars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RF Pixel handpiece treatment (Other): There is only one arm, and that is a treatment arm. For patients with wrinkles and acne scars, they are being treated with the RF Pixel handpiece to decrease the appearance of these cosmetic deficiencies. The improvement is documented in before and after photographs.
  Interventions: Device: Alma Lasers Accent RF Pixel handpiece

INTERVENTIONS:
Device: Alma Lasers Accent RF Pixel handpiece — Treatment with fractionated RF Pixel device

SUMMARY:
To assess the safety and efficacy of the Pixel RF (fractional radio frequency) module in the treatment of acne scars and wrinkles.

DETAILED DESCRIPTION:
The study design will be a prospective open label study. Up to 20 subjects of both genders with acne scars and/or wrinkles in the face will be recruited. The subjects will be treated once on clean acne scarred skin and three times on the the wrinkled skin with the Pixel RF handpiece. Each treatment duration will be approximately 30 minutes. The initial power and number of passes parameters shall be set according to the clinical indication and skin type of the subject treated (as well as the results of test sites).

Clinical improvement will be assessed by the investigator physician from the visual appearance of the treated area according to the following scale: -1 for exacerbation, 0 no change, 1 for 1%-25% improvement, 2 for 25%-50% improvement, 3 for 50%-75% improvement, and 4 for 75%-99% improvement. Adverse side effects will be scored by clinical evaluation of erythema, edema, and burns. Real-time assessments will be made as well by the investigators. Treatment and results will be documented in a Case Report Form and follow-up sessions (1, 5 days after the treatment and 1 month and 3 months after the treatment).

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting the following inclusion criteria may participate:

  * Male or female subject 18-60 years of age.
  * Clinically documented rolling and boxcar acne scars and/or wrinkles score of 2 or 3 per the Rao-Goldman scale (see section 6.5.1 for wrinkle classification).
  * Limitation to acne scared and wrinkles area: face.
  * Patients must commit to all follow-up visits.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from participation:

* Bacterial or viral infection
* Impaired immune system
* Isotretinoin (Accutane, Amnesteem, Claravis, and Sotret) in the past 6 months
* Scleroderma
* Extensive radiation therapy
* Burns in the treatment area
* Poor healing in the treatment area
* Metal implants near the treatment area
* Implantable pacemaker or automatic defibrillator/cardioverter (AICD)
* Ablative/non-ablative cosmetic intervention (deep peeling) in the past 3 months in the areas to be treated
* Active cancer
* Active collagen or vascular disease
* Pregnancy or IVF procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Improvement in the appearance of wrinkles and acne scars | 3 months
  Visual assessment of the improvement in the appearance of wrinkles and acne scars after treatment with fractionated RF.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Metropolitan MD, Glenview, Illinois
  - Dr. Zimmerman, Las Vegas, Nevada
  - Victoria Cirillo-Hyland, Bryn Mawr, Pennsylvania